CLINICAL TRIAL: NCT07156422
Title: Pathophysiological Study of the Sensitive Scalp
Acronym: SENSISCALP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC24.0318 - SENSISCALP
Record Dates: First submitted 2025-03-18; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Sensitive Scalp
Keywords: sensitive scalp

STUDY DESIGN:
Intervention Model Description: case-control study
Masking Description: Histological and innervation analyses will be carried out in a blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case group (patient with sensitive scalp) (Other): A 'sensitive scalp' group, with an overall 3S score ≥3 and a pruritus sub-score ≥2. As pruritus is widely described as the main symptom of sensitive scalp, recruitment will be based on the presence of pruritus.
  Interventions: Procedure: A scalp biopsy using a 4 mm punch in the retroauricular hair zone; Other: a general health questionnaire; Other: Questionnaires concerning their sensitive scalp
- Control group (patient with "normal" scalp) (Other): - A 'non-sensitive scalp' group, with a 3S score of 0.
  Interventions: Procedure: A scalp biopsy using a 4 mm punch in the retroauricular hair zone; Other: a general health questionnaire

INTERVENTIONS:
Procedure: A scalp biopsy using a 4 mm punch in the retroauricular hair zone — a scalp biopsy using a 4 mm punch in the retroauricular hair zone under local anesthesia
Other: a general health questionnaire — a general health questionnaire : demographics, history, treatment, smoking, alcohol consumption, phototype.
Other: Questionnaires concerning their sensitive scalp — * The characteristics of a sensitive scalp (location, chronicity, triggering and soothing factors, use of cosmetics, etc.)
  * Sensitive Scalp Score (3S)
  * Impact on quality of life: BoSS questionnaire
  * Impact of pruritus on quality of life (ItchyQol)
  Arms: Case group (patient with sensitive scalp)

SUMMARY:
Sensitive skin is defined as a syndrome manifested by the occurrence of unpleasant sensations (tingling, burning, pain, pins and needles) in response to stimuli that should not normally cause them. These unpleasant sensations cannot be explained by lesions attributable to a specific skin disease. Sensitive skin can affect different parts of the body. The scalp is a site that is often affected, with specificity linked in particular to the presence of hair and different triggering factors (styling habits, wearing of head coverings, application of cosmetics to the scalp, etc.). Sensitive scalp affects around half the population, and can have an impact on the quality of life of sufferers, particularly those whose symptoms are very intense. Women are more likely than men to have a sensitive scalp, so in order to have a more homogenous study population, we chose to include 40 women. The pathophysiology of sensitive skin is imperfectly understood, and studies specific to the sensitive scalp are very rare. However, the pathophysiology of the sensitive scalp could be different because it is a hairy area, more innervated, and less exposed to environmental factors.

DETAILED DESCRIPTION:
Each patiente will have a sample taken in the dermatology department:

* 1 skin biopsy of the scalp (non-routine medical procedure)
* Completion of questionnaires

  40 adult women
* 20 women with a sensitive scalp (cases)
* 20 women without a sensitive scalp (controls)

Patientes with the sensitive scalp will be recruited from the dermatology department. There will be no further visits, so the duration of the study is 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Adult women without dermatosis
* Collection of free and informed consent
* patient affiliated to a social security scheme

For the control group: Sensiscalp score = 0/20 Sensitive scalp group: Sensiscalp score ≥ 3/20 with pruritus sensation ≥ 2/20

Exclusion Criteria:

* Refusal to take part in the study
* Dermatosis of the scalp (psoriasis, seborrhoeic dermatitis, etc.)
* Pregnant and breast-feeding women
* Women under legal protection (guardianship, curatorship)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women are more likely than men to have a sensitive scalp, so in order to have a more homogenous study population, we chose to include 40 women.
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Study the pathophysiology of the sensitive scalp based on a study of the genes expressed in the cutaneous tissue | 1 day
  1. mRNA in biopsy by bulk transcriptomic -> Identify differentially expressed genes between the two groups (sensitive scalp and non-sensitive scalp)
  2. mRNA in biopsy by RNAscope -> Quantify and localized expression of interest's genes

SECONDARY OUTCOMES:
Histological study of skin tissue | 1 day
  1. Histological features in biopsies - Routine staining -> Visualize/Compare skin architecture between the 2 groups (sensitive scalp and non-sensitive scalp),
  2. Protein expression in biopsies - immunofluorescent staining -> Compare the status of keratinocytes between the two groups (sensitive scalp and non-sensitive scalp)
  3. Protein expression in biopsies - immunofluorescent staining -> Compare the Receptors and ion channels expression known to be involved in pruritus between the 2 groups (sensitive scalp and non-sensitive scalp)
Study of innervation | 1 day
  1) Protein expression in biopsies - immunofluorescent staining -> Quantify free nerve endings in the epidermis and the dermis and compare between the 2 groups (sensitive scalp and non-sensitive scalp)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.